CLINICAL TRIAL: NCT00866970
Title: A Phase II Study to Determine the Safety, Efficacy, and Pharmacokinetics of Multiple Intravenous Doses of ALD518 80 mg, 160 mg, and 320 mg Versus Placebo Administered to Patients With Non-Small Cell Lung Cancer-Related Fatigue and Cachexia
Brief Title: Safety, Efficacy and Pharmacokinetics of ALD518 in Patients With Non-Small Cell Lung Cancer-related Fatigue and Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALD518-CLIN-004
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2017-09

CONDITIONS: NSCLC; Fatigue; Cachexia
Keywords: Lung Cancer; Fatigue; Cachexia
MeSH Terms: conditions — Fatigue; Cachexia; Lung Neoplasms | interventions — clazakizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 (Experimental): ALD518
  Interventions: Biological: ALD518
- 2 (Experimental): ALD518
  Interventions: Biological: ALD518
- 3 (Experimental): ALD518
  Interventions: Biological: ALD518
- 4 (Placebo Comparator): No ALD518
  Interventions: Biological: Infusion of 0.9% Saline without ALD518

INTERVENTIONS:
Biological: ALD518 — ALD518 80 mg on Day 1, Week 8 and Week 16
  Arms: 1
Biological: ALD518 — ALD518 160 mg IV on Day 1, Week 8 and Week 16
  Arms: 2
Biological: ALD518 — ALD518 360 mg IV on Day 1, Week 8, and Week 16
  Arms: 3
Biological: Infusion of 0.9% Saline without ALD518 — Infusion of 0.9% Saline without addition of ALD518
  Arms: 4

SUMMARY:
The purpose of this study is to asses the safety and efficacy of ALD518 in patients with Non-Small Cell Lung Cancer-Related Fatigue and cachexia (weight-loss).

DETAILED DESCRIPTION:
This is a phase II, double-blind, randomized, placebo-controlled study of ALD518 in patients with NSCLC related fatigue and cachexia.

It is estimated that a total of 120 patients will be randomized to ALD518 80 mg, 160 mg, 320 mg, or placebo in a 1:1:1:1 ratio.

A total of eight visits (excluding the Screening visit) will take place over a period of 24 weeks: Day 1, Weeks 2, 4, 8, 12, 16, 20, and 24.

Enrolled patients will be screened within a 4 week period (Day 35 to 7). Randomization to treatment will be within a 12 day period (Day 14 to 3), before initial dosing on Day 1.

Patients will receive treatment eight weeks apart (on Day 1, and Weeks 8 and 16). All patients will remain at the clinic for at least 4 hours from the time the infusion is started. Follow-up visits will occur four and eight weeks after the last dose of study drug, at Weeks 20 and 24, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of NSCLC incurable by other treatments including surgery
* A ≥5 % loss of body weight in the preceding 3 months
* A C-reactive protein (CRP) concentration ≥ 10 mg/L
* Life Expectancy of at least 12 weeks

Exclusion Criteria:

* Treatment with chemotherapy, large-field radiotherapy, or surgery for treatment of cancer in the past 30 days
* AST/ALT ≥ 3 x ULN at screening
* Hemoglobin < 8 g/dL at Screening
* History of or active diagnosis of Tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in Safety parameters. | 20 weeks

SECONDARY OUTCOMES:
Time to symptomatic progressions at Weeks 12 and 24 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey TL Smith, MD FRCP, Study Director — Alder Biopharmaceuticals, Inc.
Locations (43):
- Australia (4):
  - Rivercity Hospital Research Centre, Auchenflower, Queensland
  - Australian Clinical Research Organisation, Kippa-Ring, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Palliative Care Launceston General Hospital, Launceston, Tasmania
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - McGill University, Department of Oncology, Montreal, Quebec
- Georgia (3):
  - A. Gvamichava National Cancer Centre, Tbilisi
  - Union Cancer Prevention Centre, Tbilisi
  - Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi
- India (13):
  - Indira Gandhi Institute of Medical Sciences, Patna, Bihar
  - Dr. Kamakshi Memorial Hospital, Pallikaranai, Chennai
  - GKNM Hospital, Pappanaickenpalayam, Coimbatore
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Kidwai Memorial Institute of Oncology, Bangalore
  - Kailash Cancer Hospital and Research Centre, Gujarat
  - IndoAmerican Cancer Institute & Research Center, Hyderabad
  - SEAROC Cancer Centre, Jaipur
  - Orchid Nursing Home, Kolkata
  - Tata Memorial Hospital, Mumbai
  - Shatabdi Hospital, Mumbai
  - Mahavir Cancer Sansthan, Patna
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune
- P3 Research LTD, Tauranga, New Zealand
- Poland (4):
  - Oddzial Chorob Pluc i Leczenia Raka Pluc, Bydgoszcz
  - Oddzial Chemioterapii Szpital Morski, Gdynia
  - II Oddzia Chorob Pluc z Pododdzialem Chemioterapii, Krakow
  - Oddzial II Chemioterapii Specjalistyczny Szpital, Szczecin
- Romania (4):
  - Professor Dr. Al Trestioreanu Institute, Bucharest
  - Professor Dr. I Chiricuta Institute of Oncology and Radiotherapy, Cluj-Napoca
  - Oradea Clinical County Hospital Medical Oncology Department, Oradea
  - County Hospital Sibiu Medical Oncology Department, Sibiu
- Russia (7):
  - Republic Oncology Dispensary, Ufa, Bashkortostan Republic
  - Territorial Clinical Oncology Dispensary, Krasnodar, Krasnodar Territory
  - Stavropol Territorial Clinical, Pyatigorsk, Stavropol Territory
  - City Clinical Hospital No. 1, Novosibirsk
  - Saint-Petersburg State Medical University, I.P. Pavlov, Saint Petersburg
  - St. Petersburg City Oncology Dispensary, Saint Petersburg
  - Yaroslavl Regional clinical Oncology Hospital, Yaroslavl
- Serbia (4):
  - Institute of Lung Diseases and TB, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Centre Kragujevac, Kragujevac
  - Institute for Pulmonary diseases of Vojvodina, Sremska